CLINICAL TRIAL: NCT03812289
Title: A Pilot Study to Assess Feasibility of Hypofractionation and Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma Patients Awaiting Liver Transplantation
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Liver Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Radiation Oncology Institute (Unknown); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Nima Nabavizadeh, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018810; NCI-2018-02864 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-18142-L; STUDY00018810 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo SBRT on days 1, 3, 5, 7, and 9 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This trial studies how well stereotactic body radiation therapy works in treating patients with liver cancer. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the use of stereotactic body radiation therapy (SBRT) in hepatocellular carcinoma (HCC) patients with advanced liver cirrhosis as a feasible approach to providing localized disease control that adequately suffices liver transplant eligibility criteria.

SECONDARY OBJECTIVE:

I. Assess preliminary efficacy and toxicity in HCC patients with advanced cirrhosis following liver SBRT.

EXPLORATORY OBJECTIVE:

I. Assess qualify of life in HCC patients with advanced cirrhosis following liver SBRT.

OUTLINE:

Patients undergo SBRT on days 1, 3, 5, 7, and 9 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 weeks, then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Must be listed or recommended to be listed for orthotopic liver transplantation at the participating institution
* Have a Child-Pugh (CP) score >= B8
* Eastern Clinical Oncology Group (ECOG) performance status =< 2, or Karnofsky performance scale > 60
* Must have a life expectancy > 12 weeks
* Safe radiation treatment planning parameters that adhere to all organs at risk constraints per section 5.1 of the protocol. If normal organs at risk constraints (including at least 700cc of uninvolved liver) are unable to be met at the lowest dose modification (30 Gy in 5 fractions), the patient is deemed ineligible for SBRT and deemed a screen failure
* Except for prior radiotherapy or radioembolization, other prior therapies to previously treated lesions, are permitted
* People of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of SBRT. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause

  * Note: Abstinence is acceptable if this is the preferred contraception for the participant
* No other prior invasive malignancy is allowed except for the following: adequately treated basal (or squamous cell) skin cancer, in situ breast or cervical cancer. Stage I or II invasive cancer treated with a curative intent without evidence of disease recurrence for at least five years

Exclusion Criteria:

* Participants have any one of the following liver tumor characteristics:

  * Have > 5 liver tumors, or
  * Maximal diameter > 5 cm
* Complete obstruction of portal venous flow to the segment of liver that includes the target lesion
* Prior radiotherapy to the upper abdomen or radioembolization of the liver, or prior thermal ablation to the target lesion
* For fiducial marker placement:

  * Have a gold allergy
  * Any coagulopathy preventing safe fiducial placement
* Contraindication to both contrast enhanced magnetic resonance imaging (MRI) and contrast enhanced computed tomography (CT) (i.e. unable to undergo follow-up imaging or SBRT treatment planning)
* Participation in another concurrent treatment protocol
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nima Nabavizadeh, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (SBRT): Patients undergo Stereotactic Body Radiation Therapy (SBRT), with 5 fractions planned for study days 1, 3, 5, 7, and 9, and a total dose of 40, 35, or 30 gray depending on normal organ constraints being met.
Period: Overall Study
Arm/Group | Treatment (SBRT)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants] — Age at study enrollment
  Participants
    <=18 years | 0
    Between 18 and 65 years | 6
    >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] — Age at study enrollment
  years | 58 [48 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Are Transplant Eligible 1 Year Following SBRT
Description: "Transplant eligible" means transplanted within 1 year or having localized disease control that meets Milan criteria at 1-year post-SBRT. Reported with 95% exact confidence interval.
Time Frame: From first SBRT dose to time of disease progression, transplantation, or 1 year after last SBRT dose (Day 374), whichever occurs first
Population: Efficacy analysis set, comprising participants who have received at least 85% of the prescribed SBRT dose
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
percentage of participants | 66.7 [29.9 to 92.5]

2. Secondary Outcome: Localized Control Rate
Description: Local control is defined as the absence of progressive disease within or at the planning target volume (PTV) margin.
Time Frame: From first SBRT dose to time of disease progression, transplantation, death, or 2 years after last SBRT dose (Day 739), whichever occurs first
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
percentage of participants | 100.0 [66.4 to 100.0]

3. Secondary Outcome: Incidence of Intrahepatic Progressive Disease
Description: Intrahepatic progressive disease is defined as development of intrahepatic recurrent or new disease within any section of the liver, including the PTV.
Time Frame: From first SBRT dose to time of intrahepatic disease progression, transplantation, death, or 2 years after last SBRT dose (Day 739), whichever occurs first.
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (SBRT): Patients undergo SBRT, with 5 fractions planned for study days 1, 3, 5, 7, and 9, and a total dose of 40, 35, or 30 gray depending on normal organ constraints being met.
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
percentage of participants | 0.0 [0.0 to 33.6]

4. Secondary Outcome: Incidence of Extrahepatic Progressive Disease
Description: Extrahepatic progressive disease is defined as progressive disease outside of the liver.
Time Frame: From first dose of SBRT to time of extrahepatic disease progression, transplantation, death, or 2 years after last SBRT dose (Day 739), whichever occurs first.
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
percentage of participants | 0.0 [0.0 to 33.6]

5. Secondary Outcome: Proportion of Participants That Proceed to Transplantation
Description: Measured and reported with 95% confidence interval.
Time Frame: as for outcome 2
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
percentage of participants | 66.7 [29.9 to 92.5]

6. Secondary Outcome: Overall Survival
Description: Reported with median survival and 95% confidence interval, if available.
Time Frame: From first SBRT dose to time of death or 2 years after last SBRT dose (Day 739), whichever occurs first.
Population: Efficacy analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
months | 13.7 [4.1 to NA] — Upper bound for 95% confidence interval was not estimable due to an insufficient number of participants with death events.

7. Secondary Outcome: Incidence of Non-classic Radiation-induced Liver Disease (RILD)
Description: Non-classic RILD is defined as grade 4 aspartate aminotransferase or alanine aminotransferase elevation, or an increase in Child-Pugh score of ≥ 2 within 1 week to 3 months after completing SBRT. Will be estimated along with an exact confidence interval.
Time Frame: From first SBRT dose to 3 months after last SBRT dose (Day 100)
Population: Safety analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
percentage of participants | 0.0 [0.0 to 33.6]

8. Secondary Outcome: Incidence of Liver Toxicity Within 1 Week to 3 Months After SBRT.
Description: Liver toxicity is assessed per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be estimated along with an exact confidence interval.
Time Frame: From 1 week (Day 16) to 3 months (Day 100) after completing SBRT
Population: Safety analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (SBRT)
Number analyzed (Participants) | 9
percentage of participants | 11.1 [0.3 to 48.2]

9. Other Pre Specified Outcome: Quality of Life (QoL) Scores for European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 Questionnaire
Description: Summary of QoL over time. No hypothesis testing is planned for QoL.
Time Frame: From screening to death or 2 years after last SBRT dose, whichever occurs first.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: QoL Scores for Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) Questionnaire
Description: Summary of QoL over time. No hypothesis testing is planned for QoL.
Time Frame: From screening to death or 2 years after last SBRT dose, whichever occurs first.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Proportion With Histopathologic Changes in Irradiated Tumor Sites Relative to Uninvolved Liver Tissue
Description: Descriptive statistical analysis of the proportion of efficacy set participants with histopathologic changes in irradiated tumor sites (of explanted livers) relative to uninvolved liver tissue.
Time Frame: At transplantation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed for up to 3.5 months. However, All-Cause Mortality was assessed for up to Day 739 (2 years after last SBRT dose).
Description: AEs will be evaluated and graded per NCI CTCAE v5.0 from the time the participant signs the consent form to 3 months following SBRT.
Arm/Group | Treatment (SBRT)
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SBRT) (N=9)
Encephalopathy (Nervous system disorders) | 2 (3)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (SBRT) (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT03812289/Prot_SAP_000.pdf